CLINICAL TRIAL: NCT04379492
Title: Single-center, Phase II, Randomized Double-blind, Placebo-controlled Study of Hydroxychloroquine Compared to Placebo as Treatment for Severe Acute Respiratory Syndrome Coronavirus 2 (SARS-CoV-2) Infection
Brief Title: A Study of Hydroxycholoroquine Compared to Placebo as Treatment for People With COVID-19
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Emerging evidence does not support the use of HCQ for treatment or prevention of SARS -CoV2 infection. No pts have been enrolled.
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 20-187
Record Dates: First submitted 2020-05-05; First posted 2020-05-07 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2020-10

CONDITIONS: COVID-19; COVID19; Sars-CoV2; SARS-Cov-2
Keywords: Sars-CoV2; SARS-Cov-2; COVID-19; COVID19; Hydroxycholoroquine; Memorial Sloan Kettering Cancer Center; 20-187
MeSH Terms: conditions — COVID-19 | interventions — Hydroxychloroquine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm A - hydroxycholoroquine (Experimental): Participants will receive hydroxycholoroquine (200-mg tablets) 2 tablets orally q12h for 2 doses on day 1 (load), followed by 1 tablet orally q12h for days 2-5.
  Interventions: Drug: Hydroxychloroquine
- Arm B - placebo (Placebo Comparator): Participants will receive placebo
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Hydroxychloroquine — Participants will receive hydroxycholoroquine (200-mg tablets) 2 tablets orally q12h for 2 doses on day 1 (load), followed by 1 tablet orally q12h for days 2-5.
  Arms: Arm A - hydroxycholoroquine
Other: Placebo — Participants will receive masked placebo given as 2 tablets orally q12h for 2 doses on day 1, followed by 1 tablet orally q12h for days 2-5.
  Arms: Arm B - placebo

SUMMARY:
This study is being done to see if hydroxychloroquine is an effective treatment for COVID-19.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years and older
* Subjects must have a documented positive test for the SARS-CoV-2 infection within 7 days of randomization
* Subject must be hospitalized within 72 hours of randomization
* Subjects must be receiving standard of care for SARS-CoV-2
* Subject/Legally Authorized Representative (LAR) must have the ability to understand and give informed consent
* Subject must be able to take and absorb hydroxychloroquine at the discretion of the investigator

Exclusion Criteria:

* Prior receipt of hydroxychloroquine for treatment or prophylaxis of SARS-CoV-2 or patient is taking hydroxychloroquine for other approved indications (e.g., lupus, rheumatoid arthritis)
* No documented SARS-CoV-2 infection
* Mechanical ventilation
* Known hypersensitivity to hydroxychloroquine or 4-aminoquinoline derivatives Preexisting retinopathy documented in medical history
* Pregnancy or Breastfeeding
* Concurrent use of any other quinine derivative (chloroquine, mefloquine) or rifamycins (rifampin, rifabutin)
* Antiarrhythmic medications (amiodarone, sotalol, dofetilide, procainamide, quinidine, flecainide)
* History of glucose-6-phosphate dehydrogenase deficiency
* Pre-treatment corrected QT interval (QTc) >500 milliseconds
* Pressor requirement to maintain blood pressure
* Alanine aminotransferase (ALT) and/or asparate aminotransferase (AST) level > 5X upper limit of normal
* Creatinine clearance <30 mL/min or requirement of dialysis or continuous venovenous hemofiltration
* Concomitant participation in a therapeutic trial for SARS-CoV-2 or receiving any experimental treatment for SARS-CoV-2 within 7 days of randomization
* Any condition that in the opinion of the principal investigator would prevent participation in the trial or would interfere with the trial endpoints

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-05-05 (Actual); Primary Completion 2020-09-25 (Actual); Study Completion 2020-09-25 (Actual)

PRIMARY OUTCOMES:
Clinical improvement on the Ordinal Scale for Clinical Improvement (OSCI) | 14 days
  Clinical improvement is defined as a composite endpoint of a two-point clinical improvement on the Ordinal Scale for Clinical Improvement (OSCI). The OSCI is an ordinal scale of 9 severity levels (from 0 to 8) for COVID-19
Number of participants requiring mechanical ventilation for respiratory failure | 14 days
  Clinical improvement is defined as no mechanical ventilation for respiratory failure attributed to SARS-CoV-2 within 14 days of randomization.

CONTACTS AND LOCATIONS:
Overall Officials: Genovefa Papanicolaou, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan - Kettering Cancer Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org